CLINICAL TRIAL: NCT01922713
Title: Effect of Daily Consumption of β-carotene Biofortified Maize on Milk Retinol Concentration in Lactating Zambian Women
Brief Title: Effect of Daily Consumption of Orange Maize on Breast Milk Retinol in Lactating Zambian Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Johns Hopkins University (Other); Tropical Diseases Research Centre, Zambia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: HP-8282
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Vitamin A Deficiency
Keywords: biofortification; vitamin A; maize; beta-carotene; breastmilk; Zambia
MeSH Terms: conditions — Vitamin A Deficiency; Callosities | interventions — Vitamin A; retinol palmitate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- white maize (Placebo Comparator): white maize and a corn oil capsule
  Interventions: Other: white maize and a corn oil capsule
- orange maize (Experimental): orange maize and a corn oil capsule
  Interventions: Other: orange maize and a corn oil capsule
- vitamin A (Active Comparator): white maize and a vitamin A capsule
  Interventions: Other: white maize and a vitamin A capsule

INTERVENTIONS:
Other: white maize and a corn oil capsule — ~ 0 ug RAE/d
  Arms: white maize
Other: orange maize and a corn oil capsule — ~600 ug RAE/d
  Other Names: beta-carotene biofortified maize
  Arms: orange maize
Other: white maize and a vitamin A capsule — 600 ug RAE/d
  Other Names: retinyl palmitate capsule
  Arms: vitamin A

SUMMARY:
The purpose of the study is to determine whether daily consumption of beta-carotene biofortified maize will increase breast milk retinol concentration in lactating Zambian women.

DETAILED DESCRIPTION:
Lactating women were randomly assigned to one of three intervention groups to receive 6d/wk for 3 wk either 1) provitamin A biofortified orange maize and a corn oil capsule, 2) white maize and a vitamin A capsule, or 3) white maize and a corn oil capsule. The 'orange maize' and 'vitamin A' groups received ~600 ug RAE/d as provitamin A biofortified maize or retinyl palmitate, respectively. The 'white maize' group was a negative control group that did not receive any supplemental vitamin A.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy lactating women 18-35 years of age
* who are breastfeeding a single infant, 4-12 mo of age.

Exclusion Criteria:

* Pregnancy,
* Chronic disease,
* Hb concentration <90 g/L,
* Signs or symptoms of vitamin A deficiency

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 149 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Breast milk retinol concentration | After 3 weeks of intervention
  Breast milk retinol concentration will be measured before and after 3 wk of consumption of orange maize (6 d/wk)

SECONDARY OUTCOMES:
Breastmilk beta-carotene concentration | After 3 wk of intervention
  Breastmilk beta-carotene concentration will be measured before and after 3 wk of consumption of orange maize (6d/wk)

OTHER OUTCOMES:
Plasma retinol concentration | After 3 wk of intervention
  Plasma retinol concentration will be measured before and after 3 wk of consumption of orange maize (6d/wk)

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie Haskell, PhD, Principal Investigator — University of California, Davis
Locations (1):
- Center for Human Nutrition, Mkushi, Mkushi District, Zambia

REFERENCES:
- [Derived] Palmer AC, Chileshe J, Hall AG, Barffour MA, Molobeka N, West KP Jr, Haskell MJ. Short-Term Daily Consumption of Provitamin A Carotenoid-Biofortified Maize Has Limited Impact on Breast Milk Retinol Concentrations in Zambian Women Enrolled in a Randomized Controlled Feeding Trial. J Nutr. 2016 Sep;146(9):1783-92. doi: 10.3945/jn.116.233700. Epub 2016 Jul 27. PMID 27466608